CLINICAL TRIAL: NCT05859711
Title: Effectiveness of Thyme Honey in Management of Xerostomia in Post Radiation Cancer Patients A Randomized Controlled Clinical Trial With a Biochemical Assessment
Brief Title: Effectiveness of Thyme Honey in Management of Xerostomia in Post Radiation Cancer Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dina Magdi, teaching assistant of oral medicine and periodontology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDASU-REC 111
Record Dates: First submitted 2023-04-05; First posted 2023-05-16 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Head and Neck Cancer Patients
Keywords: xerostomia; thyme honey; nitric oxide
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- thyme honey (Experimental): oral rinses (20 ml of thyme honey diluted in 100 ml of purified water) 3 times per day starting in the 4th week of radiotherapy and for one month after completion of radiotherapy. (Charalambous et al.,2017)
  Interventions: Drug: thyme honey mouth rinse
- Saline (Active Comparator): oral rinses with saline 3 times per day starting in the 4th week of radiotherapy and for one month after completion of radiotherapy.
  Interventions: Drug: saline mouth rinse

INTERVENTIONS:
Drug: thyme honey mouth rinse — oral rinses (20 ml of thyme honey diluted in 100 ml of purified water) 3 times per day starting in the 4th week of radiotherapy and for one month after completion of radiotherapy. (Charalambous et al.,2017)
  Arms: thyme honey
Drug: saline mouth rinse — saline mouth rinse 3 times per day starting in the 4th week of radiotherapy and for one month after completion of radiotherapy
  Arms: Saline

SUMMARY:
Xerostomia is the most frequent complication among patients who receive radiotherapy (RT) . The prevalence of xerostomia has been reported to be from 73.5% to 93% (Kakoei S.,2012). Damage to normal tissues can result by radiotherapy as it is not selective to cancer cells, and so affecting the quality of life of patients. Honey is one of the methods studied by CIM for management of HNC treatment side effects due to its properties. (Brennan et al., 2002; Clarkson et al., 2007; Furness et al., 2011;Hackett et al., 2015).

Thyme honey is a new alternative for management of xerostomia, which is a propolis gel product. Thyme honey is a variety of monofloral honey made from the nectar and pollen of thyme flowers. It has a strong antioxidant, antibacterial, antifungal and immuno modulating health effects. Due to the high sugar concentration in honey, it is believed that its presence in the oral cavity has a sialogogue effect, stimulating the salivary glands to produce saliva.

DETAILED DESCRIPTION:
90 post radiation cancer patients were randomly assigned into two equal groups.The intervention group will have oral rinses (20 ml of thyme honey diluted in 100 ml of purified water) 3 times per day starting in the 4th week of radiotherapy and for one month after completion of radiotherapy. Patients in the control arm followed the same protocol with normal saline rinses. The treatment assessment of subjective dry mouth score, objective dry mouth score, salivary Ph and salivary flow rate will be carried out at baseline, 2 weeks and one month after starting of the treatment protocol (Charalambous et al., 2017).

Nitric oxide levels will be measured at baseline and after one month of treatment (Abadi et al., 2020).

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to non-palliative head and neck radiotherapy
* Total dose of radiation received (50-70 Gy)
* Patients with complaint of xerostomia
* Age 25-65 years old
* Objective dry mouth score from ( 2-5)
* Subjective dry mouth score from (1-4)
* Undergoing radiotherapy for at least three weeks
* Can independently complete the questionnaire

Exclusion Criteria:

* Have confirmed systemic diseases or medications associated with xerostomia
* Have a known allergy to honey
* Patients who had salivary glands removal surgery
* Patients with salivary gland diseases or malignancy
* Vulnerable groups such as pregnant females, prisoners, mentally and physically handicapped individuals.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-02-20 (Actual); Primary Completion 2021-06-20 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
subjective dry mouth score | change from baseline at 4 weeks
  Q1. Do you feel dryness in your mouth ? Q2. Do you drink liquids to help you swallow dry food? Q3. Do you feel mouth dryness when eating a meal? Q4. Does the saliva seem to be too little in your mouth? Subjects who answered confirmatively to at least one of those questions related to dry mouth will be considered as positive for oral dryness subjective complaints.

SECONDARY OUTCOMES:
objective dry mouth score | change from baseline at 4 weeks
  Objective dry mouth score:
  The patients will be examined for their signs of dry mouth including:
  (Osailan et al., 2011).
  1. pooled saliva loss
  2. stickiness of mouth mirror to buccal mucosa
  3. stringy or foamy appearance of saliva
  4. dehydration of the lips
  5. no response to parotid stimulation Calculation of Objective dry mouth scores will be according to the number of dry mouth signs observed (0-5) and patients with less than 2 score will be excluded
salivary PH | change from baseline at 4 weeks
  identification of PH according to the color of the PH paper
nitric oxide levels | change from baseline at 4 weeks
  assessment of nitric oxide levels in the salivary samples using ELISA
Salivary flow rate | change from baseline at 4 weeks
  assessing unstimulated salivary flow rate in 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Susan Seif, professor, Study Director — faculty of dentistry- Ain Shams university
Locations (1):
- faculty of dentistry- Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No